CLINICAL TRIAL: NCT03519633
Title: The Role of Deep Neuromuscular Blockade and Sugammadex in Laparoscopic Hysterectomy: A Randomized Controlled Trial
Brief Title: Role of Curarization During Anesthesia for Laparoscopic Hysterectomy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Corrado Terranova, Principal investigator, Campus Bio-Medico University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GYN LPS-CUR 2018
Record Dates: First submitted 2018-03-09; First posted 2018-05-09 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2018-04

CONDITIONS: Curarization, Postoperative Residual; Postoperative Pain Of Laparoscopic Surgery; PONV
Keywords: deep neuromuscular blockade; sugammadex; postoperative pain; laparoscopic hysterectomy
MeSH Terms: conditions — Delayed Emergence from Anesthesia; Postoperative Nausea and Vomiting; Pain, Postoperative | interventions — Sugammadex; Neostigmine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Anesthesiologists were aware of the treatment assignment, while the surgeon and surgical staff were blinded. Additionally, patients, nurses/doctors assessing outcomes, and the statistician were blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SUG (Experimental)
  Interventions: Drug: Sugammadex
- NEO (Active Comparator)
  Interventions: Drug: Neostigmine

INTERVENTIONS:
Drug: Sugammadex — Reversal of deep NMB
  Arms: SUG
Drug: Neostigmine — Reversal of moderate NMB
  Arms: NEO

SUMMARY:
The primary outcome of this study is to investigate whether deep NMB reversed with Sugammadex is superior to moderate NMB reversed with Neostigmine, in terms of overall pain in the first 48 hrs after laparoscopic hysterectomy, reversal time from NMB (TOF≥0.9) and direct and indirect costs. Additionally we will also assess: drugs consumption for pain and antiemetics (rescue dose), surgical conditions, hemodynamic and respiratory stability, operation time, anesthesia time, total amount and flow rate of CO2, insufflation time, resolution of post-operative ileus, dry mouth and PONV in the first 48 hours, patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

Age 18-75 years BMI between 16 and 40 Kg/m2 ECOG Performance Status tra 0 e 1 American Society Anesthesiologist (ASA) class 1 or 3 Able to provide informed consent to trial procedures

Exclusion Criteria:

* Age < 18 or > 75 years
* BMI <16 o > 40 Kg/m2
* ECOG Performance Status >1
* Pregnancy
* Active or recent pelvic inflammation
* Anticipated airway difficulty
* Patients with history of allergy to rocuronium, neostigmine or sugammadex
* Allergy to NSAIDs
* Previous opioids consumption for chronic pain
* Patients receiving drugs for different medical conditions, that may prolong or shorten the duration of rocuronium effect (e.g aminoglycosides, magnesium)
* Hepatic or renal failure
* Persistent coagulopathy
* Neurological or cognitive disorders
* Conversion from laparoscopic to open surgery Onset of intraoperative complications

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Overall pain in the first 24 hrs after gynecologic surgical procedures | First 48 hrs after gynecologic surgical procedures
  0-10 NRS
Recovery time (or Reversal time) from NMB (TOF≥0.9) | Recovery time (or Reversal time) from NMB (TOF≥0.9) will be measured after the administration of reversal agent at the end of the surgical procedure.
  Recovery time (or Reversal time) from NMB (TOF≥0.9), measured in minutes from to administration of reversal agent to a TOF≥0.9

CONTACTS AND LOCATIONS:
Locations (1):
- Campus Bio-medico, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No